CLINICAL TRIAL: NCT00656981
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate Safety & Efficacy of Oral Contraceptive Prep., Containing Drospirenone 3 mg/Ethinyl Estradiol 20 Mcg for 6 Treatment Cycles in Women With Moderate Acne Vulgaris
Brief Title: Evaluate Safety and Efficacy of an Oral Contraceptive (OC) Preparation Versus Placebo for 6 Treatment Cycles in Women With Moderate Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91231; 306996
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Acne Vulgaris
Keywords: Moderate Acne Vulgaris; Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — drospirenone and ethinyl estradiol combination; drospirenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: YAZ (DRSP 3 mg/EE 0.02 mg, BAY86-5300)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YAZ (DRSP 3 mg/EE 0.02 mg, BAY86-5300) — The study medication was packaged in 28-tablet blister packs. Each subject kit contained 6 blister packs plus 1 reserve blister pack.Subjects randomly assigned to the active treatment group received 24 consecutive days of hormonally active tablets (3mgDRSP/0.02mgEE) followed by 4 consecutive days of inactive tablets. The treatment period was 6 cycles (28 tablets per cycle).
  Arms: Arm 1
Drug: Placebo — The subjects randomly assigned to the placebo group received 28 inert but identical-appearing, color-matched tablets. The treatment period was 6 cycles (28 tablets per cycle)
  Arms: Arm 2

SUMMARY:
The objectives of this study were to evaluate the efficacy and safety of drospirenone 3 mg/ethinyl estradiol 0.02 mg (DRSP/EE) in comparison with placebo in female subjects with moderate acne vulgaris during 6 treatment cycles

ELIGIBILITY:
Inclusion Criteria:

* Female age 14-45, with 10 to 100 comedones (noninflammatory lesions), 10 to 50 inflammatory lesions (papules or pustules), and not more than 35 nodules (<5mm) on the face).

Exclusion Criteria:

* Standard contraindications for use of combined oral contraceptives (class label)plus
* Subjects with acne and atopia, comedonal acne or acne conglobate, sandpaper acne or acne with multiple large nodes, cysts, fistular comedones, or abscessing fistular ducts
* Use of comedogenic covering cream, comedogenic sunscreens, other sex hormone preparations or any other anti-acne therapy (eg, light therapy, oleic acids, chemical peelings, mechanical extraction of comedones)
* Acne therapy with sex hormone preparations given over 3 months or longer and proved to be unsuccessful
* Preparations that have had an acne-inducing effect, eg, iodinated or bromated drugs, tuberculostatics, lithium, Vitamin B1, B6, B12, D3, corticoids, ACTH, anabolics, quinine, disulfiram, methoxypsoralen, phenobarbital, phenytoin, trimethadione, thyroid depressants, and certain oily cosmetics

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 541 (Actual)
Dates: Start 2003-01; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Percent change in inflammatory lesion counts (including papules, pustules, and nodules), non-inflammatory lesion counts (including open and closed comedones), total lesion count, and the ISGA. | From baseline to Cycle 6.

SECONDARY OUTCOMES:
Change from baseline in count of papules | Visits 3-5
Change from baseline in count of pustules | Visits 3-5
Change from baseline in count of nodules | Visits 3-5
Change from baseline in count of open comedones | Visits 3-5
Change from baseline in count of closed comedones | Visits 3-5
Percentage of subjects classified as "improved" according to the Investigator's Overall Improvement Rating | Visits 3-5
Percentage of subjects classifying themselves as "improved" on the Subject's Overall Self-Assessment Rating | Visits 3-5

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- United States (21):
  - Mobile, Alabama
  - Kingman, Arizona
  - Encino, California
  - San Diego, California
  - Westlake Village, California
  - Castle Rock, Colorado
  - Denver, Colorado
  - Palm Springs, Florida
  - St. Petersburg, Florida
  - Venice, Florida
  - Boise, Idaho
  - Shawnee, Kansas
  - Louisville, Kentucky
  - Fridley, Minnesota
  - East Steauket, New York
  - New York, New York
  - Medford, Oregon
  - Portland, Oregon
  - Byran, Texas
  - Arlington, Virginia
  - Seattle, Washington